CLINICAL TRIAL: NCT06098339
Title: Performance Evaluation of Reusable Contact Lenses When Worn For One Month By Habitual Soft Contact Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Collaborators: Centre for Ocular Research & Education, Canada (Other)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-151
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-05

CONDITIONS: Myopia; Hyperopia
MeSH Terms: conditions — Myopia; Hyperopia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Lens A, then Lens B (Experimental): Participants wore Lens A for one month and then Lens B for one month.
  Interventions: Device: Lens A (fanfilcon A); Device: Lens B (lotrafilcon B)
- Lens B, then Lens A (Experimental): Participants wore Lens B one month and then Lens A for one month.
  Interventions: Device: Lens A (fanfilcon A); Device: Lens B (lotrafilcon B)

INTERVENTIONS:
Device: Lens A (fanfilcon A) — Daily wear for one month
Device: Lens B (lotrafilcon B) — Daily wear for one month

SUMMARY:
The purpose of this study was to compare the clinical performance of two different reusable lenses in habitual spherical soft lens wearers.

DETAILED DESCRIPTION:
This study was a prospective, bilateral eye, double-masked, randomized, 1 month cross-over, daily-wear design involving two different frequent replacement type lenses. Duration of involvement for each participant was approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

1. Were at least 18 years of age and no older than 39 years, and had full legal capacity to volunteer;
2. Had read and signed an information consent letter;
3. Were willing and able to follow instructions and maintain the appointment schedule;
4. Self-reported having had a full eye examination in the previous two years;
5. Had healthy eyes with no health condition or medication that contra-indicate contact lens wear, in the opinion of the investigator;
6. Anticipated being able to wear the study lenses for at least 8 hours a day, 6 days a week;
7. Habitually wore spherical soft contact lenses, for the past 3 months minimum:

   It was preferred that all participants were habitual frequent replacement lens wearers. However, if this was not possible then no more than 5 participants could be habitual daily disposable lens wearers at each site, the rest had to be habitual frequent replacement lens wearers;

   - For the frequent replacement wearers: No more than 3 could be habitual wearers of the Avaira Vitality™/ Serenity™ brand (or their equivalent private label brand name) and no more than 3 could be habitual wearers of AIR OPTIX® plus HydraGlyde® can be enrolled at each site;
8. Had refractive astigmatism no higher than -0.75DC in each eye;
9. Could be fit and achieve binocular distance vision of at least 20/30 Snellen (Available lens parameters are sphere +6.00 to -6.00D, 0.25D steps).

Exclusion Criteria:

1. Were participating in any concurrent clinical or research study;
2. Had any known active ocular disease and/or infection that contraindicated contact lens wear;
3. Had a systemic or ocular condition that in the opinion of the investigator may have affected a study outcome variable;
4. Were using any systemic or topical medications that in the opinion of the investigator may have affect contact lens wear or a study outcome variable;
5. Had known sensitivity to the diagnostic sodium fluorescein used in the study;
6. Self-reported as pregnant, lactating or planning a pregnancy at the time of enrolment;
7. Had undergone refractive error surgery or intraocular surgery.

Ages: 18 Years to 39 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 53 (Actual)
Dates: Start 2023-11-13 (Actual); Primary Completion 2024-04-04 (Actual); Study Completion 2024-04-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carolyn MacNeil, Principal Investigator — Insight Eye Care; Abigail Gillogly-Harsch, Principal Investigator — Nittany Eye Associates; Roxanne Achong-Coan, Principal Investigator — Coan Eye Care
Locations (3):
- United States (2):
  - Coan Eye Care, Ocoee, Florida
  - Nittany Eye Associates, State College, Pennsylvania
- Insight Eye Care, Waterloo, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Lens B, Then Lens A: Participants wore Lens B for one month and then Lens A for one month.
Period: Period 1: First Intervention 28-32 Days
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 25 | 28
Completed | 24 | 26
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Enrolled outside the study inclusion/exclusion criteria and was discontinued early | 1 | 1
Period: Period 2: Second Intervention 28-32 Days
Arm/Group | Lens A, Then Lens B | Lens B, Then Lens A
Started | 24 | 26
Completed | 24 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total Study Population: All participants that were dispensed intervention (Lens A or Lens B), regardless of eligibility or study completion
Arm/Group | Total Study Population
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Lens Handling on Removal
Description: Participants measured subjective lens handling at removal on a 0-100 integer scale, where 0=worst and 100=best. Results for each lens were collected in the at-home diary on Day 27.
Time Frame: Day 27
Population: Analysis population includes all participants that were eligible (inclusion/exclusion criteria) and completed all study visits. Of 50 participants that completed the study, 1 was removed from the analysis due to a symptomatic adverse event at the final study visit which may have impacted the study data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Lens A: Participants that received Lens A during either the first or second period of the study
- Lens B: Participants that received Lens B during either the first or second period of the study
Arm/Group | Lens A | Lens B
Number analyzed (Participants) | 49 | 49
score on a scale | 84 (21) | 89 (17)

ADVERSE EVENTS:
Time Frame: The duration of the clinical trial, approximately 2-3 months
Groups:
- Lens A: Participants that received Lens A
- Lens B: Participants that received Lens B
Arm/Group | Lens A | Lens B
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 0/50
Other Adverse Events (participants affected / at risk) | 5/50 | 4/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lens A (N=50) | Lens B (N=50)
Viral conjunctivitis (Eye disorders) | 0 (0) | 1 (2)
Ocular discomfort, (Eye disorders) | 3 (5) | 0 (0)
Asymptomatic corneal infiltrate event (Eye disorders) | 1 (1) | 1 (1)
Lower lid small chalazion (Eye disorders) | 0 (0) | 1 (1)
Nasal upper lid papilloma (Eye disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/39/NCT06098339/Prot_SAP_001.pdf